CLINICAL TRIAL: NCT03056248
Title: Lithium in Cardiac Surgery Related Acute Kidney Injury: A Pilot Study
Brief Title: Lithium in Acute Kidney Injury
Acronym: LSCAKI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lifespan (Other)
Responsible Party: Principal Investigator, Sairah Sharif, Assistant Professor, Lifespan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 02116
Record Dates: First submitted 2017-02-13; First posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Lithium Carbonate; Lithium

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to lithium versus placebo and rates of acute kidney injury will be measured
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients and investigators will be blinded to the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lithium (Active Comparator): Patients will be identified by chart review and be explained the purpose of the study and informed consent taken
  Interventions: Drug: Lithium Carbonate
- Placebo (Placebo Comparator): Patients will be identified by chart review and be explained the purpose of the study and informed consent taken
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Placebo oral capsule — On day 0, the day of the cardiac surgery placebo will be given once On day 1, one day after cardiac surgery placebo will be given once On day 2, two days after cardiac surgery placebo will be given once
  Other Names: Placebo
  Arms: Placebo
Drug: Lithium Carbonate — On day 0, the day of the cardiac surgery oral lithium will be given at dose 900mg once On day 1, one day after cardiac surgery oral lithium will be given at dose 900mg once On day 2, two days after cardiac surgery oral lithium will be given 900mg once
  Other Names: Lithium
  Arms: Lithium

SUMMARY:
A growing body of pre-clinical evidence suggests that glycogen synthase kinase 3β (GSKβ) is implicated in the development and progression of acute kidney injury (AKI). Lithium is a naturally occurring standard inhibitor of GSKβ. The purpose of this study is to examined if low dose lithium carbonate is able to reduce the incidence of AKI in patients undergoing cardiac surgery who are placed on cardiopulmonary bypass during surgery. We hypothesize that low dose lithium might reduce the incidence and duration of AKI in patients undergoing cardiac surgery who are on cardiopulmonary bypass.

DETAILED DESCRIPTION:
Cardiac surgery associated acute kidney injury (CSA-AKI) is a significant problem. The prevalence varies from 0.3% to 22.9% depending on the definition of AKI. The pathogenesis of AKI in this population is multifactorial. Factors associated with AKI in such patients include increased age, preoperative elevated creatinine, presence of diabetes, reduced ejection fraction, increased body weight, and presence of carotid artery bruit, duration of cardiopulmonary bypass, aortic cross clamp time, and duration of surgery. CSA-AKI is an independent predictor of mortality, morbidity, increased length of stay and hospitalization costs. Moreover these patients are also at increased risk of chronic kidney disease and end stage renal failure in the future.

Various pharmacologic approaches that have been tried to prevent early CSA-AKI such as diuretics, vasodilators, and anti-inflammatory drugs. Fenoldopam, atrial natriuretic peptide, and brain natriuretic peptide have shown little renoprotection. However these strategies lack high quality evidence to support their use and are not standard of care. There is no strong evidence to suggest any single or multiple pharmacotherapy that significantly impacts in reducing CAS-AKI. Thus the current best therapy for CSA-AKI is prevention, supportive care, hemodynamic optimization and renal replacement therapy.

AKI is an extremely complex process involving multiple pathophysiologic pathways. Glycogen synthase kinase 3β (GSK3β) is implicated in many pathways beyond glycogen metabolism and has been shown to be an important player in the development of AKI . Lithium is a US Food and Drug Administration (FDA)-approved drug which has been used for over 50 years as first line agent to treat mood disorders. It is a standard inhibitor for GSK3β. Latest evidence in murine models of cisplatin-induced AKI and ischemia/reperfusion-induced AKI suggests that lithium treatment may attenuated kidney dysfunction and kidney histologic injury following AKI. Lithium was able to promote kidney tubular cell repair hence improvement of AKI in murine models. In addition, lithium has also been found to exert an anti-proteinuric and renal reparative effect. On this background we want to explore the potential preventive and therapeutic role of lithium carbonate in CSA- AKI.

ELIGIBILITY:
Inclusion Criteria:

* A male or female greater than 18 years
* Stable renal function with creatinine change <0.3mg/dl in the preceding 1 month prior to scheduled surgery
* Procedure such as aortic valve surgery, mitral valve surgery, coronary artery bypass grafting, or combination of the above mentioned procedures
* Have estimated glomerular filtration rate greater than or equal to 15ml/min/ 1.73m2 as calculated by chronic kidney disease Epidemiology Collaboration (CKD-EPI) formula

Exclusion Criteria:

Subjects who:

* Are taking lithium prior to surgery for any reason
* Have ejection fraction of <30% prior to surgery
* Have estimated glomerular filtration rate <15ml/min/ 1.73m2 as calculated by chronic kidney disease Epidemiology Collaboration (CKD-EPI) formula
* Having cardiac surgery to be performed without using cardiopulmonary bypass
* Has ongoing sepsis or history of sepsis in the last 2 weeks, defined as having 2 of the following criteria T >38C or <36C, pulse rate >90/min, RR >20/min, WBC >12 or >10% polymorphonuclear cells plus a documented source
* Has documented rise in creatinine ≥ 0.3mg/dl in the preceding one month prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2017-12-30 (Estimated); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in serum creatinine mg/dl | 1 month
  Renal function

SECONDARY OUTCOMES:
Peak creatinine mg/dl | 1 month
  Renal function
Neutrophil gelatinase-associated lipocalcin (NGAL) ng/ml | 3 days
  Renal function
Kidney injury molecule-1 (KIM1) ng/ml | 3 days
  Renal function

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Reddy DS, Reddy MS. Serum Lithium Levels: Ideal Time for Sample Collection! Are We Doing it Right? Indian J Psychol Med. 2014 Jul;36(3):346-7. doi: 10.4103/0253-7176.135399. PMID 25035570
- [Result] Vives M, Wijeysundera D, Marczin N, Monedero P, Rao V. Cardiac surgery-associated acute kidney injury. Interact Cardiovasc Thorac Surg. 2014 May;18(5):637-45. doi: 10.1093/icvts/ivu014. Epub 2014 Feb 16. PMID 24535092
- [Result] Gammelager H, Christiansen CF, Johansen MB, Tonnesen E, Jespersen B, Sorensen HT. Five-year risk of end-stage renal disease among intensive care patients surviving dialysis-requiring acute kidney injury: a nationwide cohort study. Crit Care. 2013 Jul 22;17(4):R145. doi: 10.1186/cc12824. PMID 23876346
- [Result] Coleman MD, Shaefi S, Sladen RN. Preventing acute kidney injury after cardiac surgery. Curr Opin Anaesthesiol. 2011 Feb;24(1):70-6. doi: 10.1097/ACO.0b013e3283422ebc. PMID 21157303
- [Result] Gong R, Wang P, Dworkin L. What we need to know about the effect of lithium on the kidney. Am J Physiol Renal Physiol. 2016 Dec 1;311(6):F1168-F1171. doi: 10.1152/ajprenal.00145.2016. Epub 2016 Apr 27. PMID 27122541
- [Result] Bao H, Ge Y, Wang Z, Zhuang S, Dworkin L, Peng A, Gong R. Delayed administration of a single dose of lithium promotes recovery from AKI. J Am Soc Nephrol. 2014 Mar;25(3):488-500. doi: 10.1681/ASN.2013040350. Epub 2014 Jan 9. PMID 24408869
- [Derived] Sharif S, Chen B, Brewster P, Chen T, Dworkin L, Gong R. Rationale and Design of Assessing the Effectiveness of Short-Term Low-Dose Lithium Therapy in Averting Cardiac Surgery-Associated Acute Kidney Injury: A Randomized, Double Blinded, Placebo Controlled Pilot Trial. Front Med (Lausanne). 2021 Jun 14;8:639402. doi: 10.3389/fmed.2021.639402. eCollection 2021. PMID 34195206